CLINICAL TRIAL: NCT01322750
Title: Circulating Tumor Cells (CTCs): A Potential Screening Test for Clinically Undetectable Breast Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Bureau of Navy Medicine (BUMED) (Unknown)
Responsible Party: Thomas A Summers, Jr, Walter Reed Army Medical Center
Other Study IDs: 354344
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Breast Abnormality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With CTCs: Those individuals whom are identified with CTCs
- Without CTCs: Those individuals whom present and did not have CTCs

SUMMARY:
With an estimated > 2 million women with undetected breast cancer in the United States, the need for improved early detection is imperative. Early diagnosis for these women is key to minimizing quality life-years lost to disease and optimizing success of treatment. Evidence now exists supporting the finding that systemic spread is an early event in the natural history of breast cancer, manifested as a release of single cancer cells from the incident, clinically undetectable tumor, which circulate through the bloodstream and deposit within remote tissues. Reliable and accurate detection of these circulating tumor cells (CTCs) is now possible with a simple peripheral venous blood draw. This study hypothesizes that women with CTCs and no other signs of malignancy have clinically undetectable disease.

This study will attempt to validate this technology as a breast cancer screening test and acquire data to determine the clinical validity and utility of this proposed screening methodology on a relatively young, ethnically diverse population who are eligible military health care beneficiaries. Furthermore, this study will attempt to bank identified CTCs in order to perform additional molecular analyses in the future. The specific aims are to develop a simple, reliable, cost-effective, and clinically relevant breast cancer screening test in order to identify subclinical disease early in its natural history in subjects at risk of progression to clinically apparent disease over the ensuing decade. The ultimate goal is to decrease the treatment-related morbidity and cause-specific mortality of breast cancer. An experienced team devoted to the care of patients with breast disease has been assembled to achieve this goal.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Mentally competent and willing to provide written informed consent prior to entering the study
* Military healthcare beneficiary
* Undergoing a diagnostic or therapeutic procedure (biopsy, lumpectomy, mastectomy) in the breast clinic or operating room.
* Present to the CBCP and willing to be followed at the CBCP during the course of treatment and follow-up

Exclusion Criteria:

* Prior history of invasive carcinoma
* Presence of clinically-apparent metastatic disease
* Participants with known human immunodeficiency virus (HIV), any history of hepatitis, prion-mediated disease, drug resistant tuberculosis or other infectious disease presenting a significant risk to personnel handling tissue or blood-derived products shall be excluded from participation
* Participants with pre-existing coagulopathies or all other conditions, for whom invasive biopsy or surgery is medically contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults (> 18 years of age) presenting for evaluation at breast center - who subsequently undergo a diagnostic or therapeutic procedure and who do not have a prior history of invasive carcinoma or clinically-apparent metastatic disease, will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 3125 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-01 (Estimated); Study Completion 2023-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States